CLINICAL TRIAL: NCT04426396
Title: Coronary CT Angiography-Derived Fractional Flow Reserve for Functional Evaluation of Coronary Artery Disease
Brief Title: Diagnostic Performance of Fractional Flow Reserve Derived From Coronary CT Angiography
Acronym: ACCURATE-CT
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-375
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FFR — FFR measured by pressure wire, CT-FFR computed by coronary CT angiography
  Other Names: CT-FFR

SUMMARY:
This is a blind evaluation, self-control, multicenter clinical trial designed to determine the diagnostic performance of CT-FFR from coronary computed tomographic angiography (CCTA), as compared to CCTA alone, for non-invasive diagnosis of the presence of a hemodynamically significant coronary stenosis, using invasive fractional flow reserve (FFR) as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years old;
* Subjects with clinical need and consent for coronary angiography;
* Can provide the results of coronary CT angiography within 60 days prior to ICA or agree to undergo coronary CT angiography;
* The subjects knew about the experiment and signed the informed consent voluntarily.

Exclusion Criteria:

* Patients who have had percutaneous coronary intervention (PCI);
* Patients who had CABG;
* Acute coronary syndrome, such as acute ST segment elevation;
* Severe tachycardia or arrhythmia;
* Patients with severe hepatorenal insufficiency;
* Patients with congenital heart disease, implanted pacemaker or defibrillator, artificial heart valve;
* Failure to perform invasive FFR examination or obtain FFR value due to various reasons;
* Allergic to β - blockers, nitrates and adenosine, sick sinus syndrome, long QT syndrome, severe hypotension, severe asthma, severe COPD or COPD;
* Persistent or significant clinical instability, including acute chest pain (sudden onset), cardiogenic shock, blood pressure instability (systolic blood pressure < 90mmHg) and severe congestive heart failure (according to the heart classification of the New York Heart Association, grade III or IV of cardiac function) or acute pulmonary edema;
* The CTA images of coronary artery showed that the stenosis rate was less than 30% or greater than 90%, or the diameter of diseased segment was less than 2.0mm;
* CT-FFR can not be calculated because of the quality of CTA image;
* Known pregnant and lactating women;
* Having participated in other clinical trials within 3 months;
* Other situations that the researchers judged were not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with stable angina or unstable angina who need selective surgery referred to coronary angiography and physiological evaluation.
Sampling Method: Probability Sample
Enrollment: 339 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of CT-FFR compared to FFR | 1 day

SECONDARY OUTCOMES:
Diagnostic accuracy and AUC of CT-FFR compared to FFR | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Li C, Hu Y, Jiang J, Dong L, Sun Y, Tang L, Du C, Yin D, Jiang W, Leng X, Jiang F, Pan Y, Jiang X, Zhou Z, Koo BK, Xiang J, Wang J; ACCURATE-CT Investigators. Diagnostic Performance of Fractional Flow Reserve Derived From Coronary CT Angiography: The ACCURATE-CT Study. JACC Cardiovasc Interv. 2024 Sep 9;17(17):1980-1992. doi: 10.1016/j.jcin.2024.06.027. Epub 2024 Aug 21. PMID 39177553